CLINICAL TRIAL: NCT04496128
Title: Neurological Complications of COVID-19
Brief Title: COVID19 Neurological Manifestation
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Sherry Hsiang-Yi Chou, Associate Professor, University of Pittsburgh
Other Study IDs: STUDY20040037
Record Dates: First submitted 2020-07-13; First posted 2020-08-03 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-04

CONDITIONS: SARS-CoV 2; Neurologic Manifestations
MeSH Terms: conditions — Neurologic Manifestations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective observational cohort study to document the prevalence and types of neurological manifestations among hospitalized patients with confirmed or suspected novel coronavirus infection (COVID-19).

DETAILED DESCRIPTION:
This study is a prospective observational cohort study to document the prevalence and types of neurological manifestations among hospitalized patients with confirmed or suspected novel coronavirus infection (COVID-19). Severe acute respiratory syndrome 2 (SARS-CoV-2), the virus that causes COVID-19, shares significant structural and biological similarities with SARS-CoV, which is known to be neuroinvasive particularly with brainstem involvement. There are emerging reports of neurological symptoms associated with COVID-19 infections, including seizures, coma, encephalitis, Guillan-Barre syndrome, and cerebrovascular events including ischemic stroke, ICH, and cerebral venous sinus thromboses. However, the exact prevalence of these conditions and their impact on patient disease severity and outcomes is unknown. As the incidence and severity of COVID-19 infection continue to rapidly rise globally, it is imperative to capture prospective data to accurately document prevalence, severity and clinical characterization of neurological components of COVID 19, the influence of treatment regimens of neurological complications, and role of these confounders on patient and organizational outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than or equal to 18 years old
* Admitted with suspected or confirmed COVID19 infection
* Patient exhibiting acute neurological symptoms

Exclusion Criteria:

* Patients under the age of 18 years old
* Pre-existing, baseline severe neurologic dysfunction including baseline coma/vegetative state, baseline quadriparesis, baseline refractory seizure disorder with frequent breakthrough seizures despite anticonvulsant use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to acute care hospital who are suspected and/or confirmed to have COVID 19.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of neurological manifestations | During hospital course, up to 1 month
  Proportion of patients with neurological symptoms out of all hospitalized COVID19 patients during study period.
Hospital Mortality | At hospital discharge, approximately 1 month
Global functional outcomes using modified Rankin score | At hospital discharge, approximately 1 month
  Patients will be assessed on a scale score of 0 (no symptoms at all) to 5 (severe disability; bedridden, incontinent and requiring constant nursing care and attention)

SECONDARY OUTCOMES:
Length of ICU stay | At hospital discharge, approximately 1 month
Length of hospital stay (in days) | At hospital discharge, approximately 1 month
30-day mortality | 30 days from the first day of hospitalization
90-day mortality | 90 days from the first day of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Sherry H Chou, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Needham EJ, Chou SH, Coles AJ, Menon DK. Neurological Implications of COVID-19 Infections. Neurocrit Care. 2020 Jun;32(3):667-671. doi: 10.1007/s12028-020-00978-4. PMID 32346843
- [Background] Frontera J, Mainali S, Fink EL, Robertson CL, Schober M, Ziai W, Menon D, Kochanek PM, Suarez JI, Helbok R, McNett M, Chou SH; GCS-NeuroCOVID Study. Global Consortium Study of Neurological Dysfunction in COVID-19 (GCS-NeuroCOVID): Study Design and Rationale. Neurocrit Care. 2020 Aug;33(1):25-34. doi: 10.1007/s12028-020-00995-3. PMID 32445105